CLINICAL TRIAL: NCT05143359
Title: Accuracy of Variables for Wharfe Assessment and Pederson Difficulty Index for Impacted Mandibular Third Molar Surgery
Brief Title: Accuracy of Variables for Impacted Mandibular Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Gobind Ram, Accuracy of variables for Wharfe assessment and Pederson difficulty index for impacted mandiblar third molar surgery---A prospective clinical study, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GOBINDRAM
Record Dates: First submitted 2021-10-16; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wharfe and Pederson difficulty index (Experimental): Assessment of Difficulty in third molar extraction using Wharfe and Pederson difficulty index
  Interventions: Diagnostic Test: Wharfe and Pederson difficulty index
- Winters difficulty index (Active Comparator): Assessment of Difficulty in third molar extraction using Winters difficulty index
  Interventions: Diagnostic Test: Winters difficulty index

INTERVENTIONS:
Diagnostic Test: Wharfe and Pederson difficulty index — Efficiency of Wharfe and Pederson Difficulty index in extraction of third molars.
  Arms: Wharfe and Pederson difficulty index
Diagnostic Test: Winters difficulty index — Efficiency of Winters Difficulty index in extraction of third molars.
  Arms: Winters difficulty index

SUMMARY:
Accuracy of the variables used in Wharfe assessment and Pederson difficulty index for impacted mandibular third molar surgery.

The lower 3rd molar tooth is one of the most frequently impacted teeth. Its prevalence ranges from 30.3% to 68.6% worldwide according to a study conducted by Sekhar, 2020. The impaction of a tooth can be defined as a pathological condition in which eruption of tooth is not normal i.e. it is not erupted as expected within a specific time period. The impaction renders the affected tooth as non-functional due to its postural instability/ abnormal position. The normal tooth eruption is dependent on several local as well as systemic factors. Normal eruption can be altered by neighboring tooth, excessive soft tissue in the surrounding, or the dense overlying bone. Race and Ethnicity an also affect/ alter the impaction rate.

The removal of 3rd mandibular molar/ wisdom tooth is one of the most commonly performed surgical procedures, being done in dental clinics on daily basis. To predict the difficulty level of this procedure for impacted lower 3rd molar, no scoring system/ scale is considered sufficient i.e. every scale takes some factors into account, while missing some factors, so clinically not very much reliable. Some of the proposed scales/ models which are clinically in use are as follows: WHARFE's, Pederson's, Winter's, and Pell and Gregory's model.

DETAILED DESCRIPTION:
The lower 3rd molar tooth is one of the most frequently impacted teeth. Its prevalence ranges from 30.3% to 68.6% worldwide according to a study conducted by Sekhar, 2020.The impaction of a tooth can be defined as a pathological condition in which eruption of tooth is not normal i.e. it is not erupted as expected within a specific time period. The impaction renders the affected tooth as non-functional due to its postural instability/ abnormal position. The normal tooth eruption is dependent on several local as well as systemic factors. Normal eruption can be altered by neighboring tooth, excessive soft tissue in the surrounding, or the dense overlying bone. Race and Ethnicity an also affect/ alter the impaction rate.

The removal of 3rd mandibular molar/ wisdom tooth is one of the most commonly performed surgical procedures, being done in dental clinics on daily basis. To predict the difficulty level of this procedure for impacted lower 3rd molar, no scoring system/ scale is considered sufficient i.e. every scale takes some factors into account, while missing some factors, so clinically not very much reliable. Some of the proposed scales/ models which are clinically in use are as follows: WHARFE's, Pederson's, Winter's, and Pell and Gregory's model.

WHARFE's scoring system is a common classification/ system for the difficulty assessment while planning to remove a 3rd mandibular molar tooth. WHARFE stands for Winter's lines, Height of mandible, Angulation, Root, shape, & morphology, Follicular size, Exit pathway for tooth. This system helps to examine a tooth in more detail and its radiological status before planning any intervention to 3rd molar. While, Pederson's difficulty assessing scale is to predict the pre-operative and operative difficulty while riming the 3rd Mandibular Molar tooth that is impacted. It takes into account following variables: spatial relationship, depth, and ramus relationship. It is reported as slightly difficult (score 3-4), moderately difficult (score 5-6), and very difficult (score 7-10) with relation to the scores mentioned.

While doing research, I found that there is a handsome data available on different clinical scoring systems and their practical significance. But, I found the paucity of literature on the comparison of the variables used in Pederson's and WHARFE's scoring systems with practical procedures. So, this study was planned to assess the credibility of these variables. This study will also explore whether these systems are sufficient enough to rely upon, while (intelligently) planning intervention in the patients presenting with lower 3rd molar impaction. It will surely help to broaden the horizon of knowledge, followed by suggesting some guidelines to improve the clinical practice while treating these patients. The relevant data will be taken from participants and their relevant investigation results will be noted down in the pre-designed Performa (attached). This data will be interpreted in the SPSS version 23.0 (Statistical Package for the Social Sciences) program and will be followed by recommendations to improve the health care standards in Pakistan. This will ultimately update the knowledge and clinical approach of treating Oral & Maxillofacial Surgeons.

MATERIAL AND METHODS:

Study Design:

Observational Study Setting: The study will be conducted in the Oral & Maxillofacial Department on the patients visiting Dr Ishrat-ul-Ebad Khan Institute of Oral Health Sciences/ DUHS Karachi on outdoor basis or indoor basis.

Duration of Study:

Six months after the approval of synopsis.

Sample Size:

A total of 281 cases is calculated as sample size, from online calculator (from www.openepi.com) keeping confidence interval of 95% and the power of 80%, while taking the difficulty index as 24%, of molar teeth as 'very difficult' to operate, when Pederson scale index was applied. (Sekhar, M., Singh, S., & Valluri, R et al. Correlation of Variables for WHARFE Assessment and Pederson Difficulty Index for Impacted Mandibular Third Molar Surgery-A Prospective Clinical Study. Journal of Maxillofacial and Oral Surgery. 2020 July 25;1(1):1 -5. https://link.springer.com/article/10.1007%2Fs12663-020-01362-7)

Sampling Technique:

Purposive non-probability sampling technique would be used for the selection of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 60 years with either gender
2. Patients having impacted 3rd mandibular molar according to Winter's classification (as per operational definition)
3. Patients with no evidence of dental caries or restoration in the past

Exclusion Criteria:

1. Patients with history of orthodontic treatment or periodontal surgery
2. Patients having craniofacial anomalies, congenital deformities or syndromes
3. Patients with evidence of cyst or tumor in the molar area
4. Not willing to participate in my study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Extraction of mandibular 3rd molar | Extraction of mandibular 3rd molar assessment by Wharfe and Peterson's index immediately after the intervention/procedure/surgery
  Difficulty of extraction will be assessed by difficulty index
Extraction of mandibular 3rd molar | Extraction of mandibular 3rd molar assessment by winters immediately after the intervention/procedure/surgery
  Difficulty of extraction will be assessed by difficulty index

CONTACTS AND LOCATIONS:
Overall Officials: Gobind Ram, Principal Investigator — Dow University of Health Sciences